CLINICAL TRIAL: NCT06541262
Title: Phase I/II Study of Silmitasertib (CX-4945) in Combination With Chemotherapy in Children and Young Adults With Relapsed Refractory Solid Tumors
Brief Title: Silmitasertib (CX-4945) in Combination With Chemotherapy for Relapsed Refractory Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Giselle Sholler, Beat Childhood Cancer Chair, Milton S. Hershey Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BCC021
Record Dates: First submitted 2024-08-02; First posted 2024-08-07 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Neuroblastoma; Ewing Sarcoma; Osteosarcoma; Rhabdomyosarcoma; Liposarcoma
MeSH Terms: conditions — Neuroblastoma; Sarcoma, Ewing; Osteosarcoma; Rhabdomyosarcoma; Liposarcoma | interventions — silmitasertib; Irinotecan; Temozolomide; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase I- Dose level 1 (Experimental): Silmitasertib 600 mg/m2 twice a day plus Neuroblastoma: Regimen A: Irinotecan and Temozolomide Sarcoma: Regimen B: Vincristine, Irinotecan and Temozolomide
  Interventions: Drug: Silmitasertib; Drug: Irinotecan; Drug: Temozolomide; Drug: Vincristine
- Phase I- Dose level 2 (Experimental): Silmitasertib 800 mg/m2 twice a day plus Neuroblastoma: Regimen A: Irinotecan and Temozolomide Sarcoma: Regimen B: Vincristine, Irinotecan and Temozolomide
  Interventions: Drug: Silmitasertib; Drug: Irinotecan; Drug: Temozolomide; Drug: Vincristine
- Phase II- Relapsed/refractory Neuroblastoma (Experimental): Silmitasertib RP2D twice a day plus Irinotecan and Temozolomide
  Interventions: Drug: Silmitasertib; Drug: Irinotecan; Drug: Temozolomide
- Phase II- Relapsed/refractory Ewing sarcoma (Experimental): Silmitasertib RP2D twice a day plus Vincristine, irinotecan and temozolomide
  Interventions: Drug: Silmitasertib; Drug: Irinotecan; Drug: Temozolomide; Drug: Vincristine

INTERVENTIONS:
Drug: Silmitasertib — Capsules
  Other Names: CX-4945
Drug: Irinotecan — IV
Drug: Temozolomide — Oral
Drug: Vincristine — IV
  Arms: Phase I- Dose level 1; Phase I- Dose level 2; Phase II- Relapsed/refractory Ewing sarcoma

SUMMARY:
The purpose of this study is to evaluate the investigational drug, silmitasertib (a pill taken by mouth), in combination with FDA approved drugs for solid tumors. An investigational drug is one that has not been approved by the U.S. Food & Drug Administration (FDA), or any other regulatory authorities around the world for use alone or in combination with any drug, for the condition or illness it is being used to treat.

The goals of this part of the study are:

* Establish a recommended dose of silmitasertib in combination with chemotherapy
* Test the safety and tolerability of silmitasertib in combination with chemotherapy in subjects with cancer
* To determine the activity of study treatments chosen based on:
* How each subject responds to the study treatment
* How long a subject lives without their disease returning/progressing

ELIGIBILITY:
Inclusion Criteria:

1. Age: Less than 30 years old at initial diagnosis
2. Pathology All subjects must have a confirmed diagnosis of tumor type. Phase I: Relapsed/refractory solid tumors: Neuroblastoma, Ewing Sarcoma, Osteosarcoma, Rhabdomyosarcoma, Liposarcoma

   Phase II:
   * Relapsed/refractory Neuroblastoma
   * Relapsed/refractory Ewing sarcoma
3. Tumor assessment:

   Disease assessment is required for eligibility and must be done after last dose of previous therapy and prior to first dose of study drug.
4. Disease Status:

   Relapsed/Refractory Neuroblastoma Relapsed disease defined as neuroblastoma that was previously in remission after standard therapy (at least 4 cycles of aggressive multi-drug induction chemotherapy, with or without radiation and surgery, followed by immunotherapy, or according to a standard high-risk treatment/neuroblastoma protocol) and has now relapsed and is in any number of relapses.

   Refractory disease defined as High-risk neuroblastoma (as defined by INRG) that failed to achieve CR after at least 4 cycles of aggressive multi-drug induction chemotherapy, progression during upfront therapy or with disease remaining after standard immunotherapy.

   International Neuroblastoma Risk Group Staging System (INRG) High Risk NB defined as one of the following:
   1. Any age with International Neuroblastoma Risk Group (INRG) Stage L2, MS, or M with MYCN amplification
   2. Age ≥ 547 days and INRG Stage M regardless of biologic features
   3. Any age initially diagnosed with INRG Stage L1 MYCN amplified NBL who have progressed to Stage M without systemic chemotherapy
   4. Age ≥ 547 days of age initially diagnosed with INRG Stage L1, L2, or MS who have progressed to Stage M without systemic chemotherapy

   Relapsed/refractory Sarcoma Subjects that have relapsed following standard of care therapy or having progressed during standard of care therapy. Standard of care therapy for sarcoma includes multi-agent chemotherapy with local control consisting of either surgery or radiation therapy.
5. Measurable or evaluable disease, including at least one of the following:

   * Measurable tumor by CT or MRI
   * MIBG or PET that is positive for disease
   * Bone Marrow biopsy/aspirate that is positive for disease
6. Timing from prior therapy:

   Subjects must have fully recovered from the acute toxic effects of all prior anti- cancer therapy and be within the following timelines:
   1. Myelosuppressive chemotherapy: Must not have received within 2 weeks of enrollment onto this study.
   2. Small Molecule Inhibitors (anti-neoplastic agent): At least 2 weeks from the completion of therapy with a small molecule inhibitor.
   3. Immunotherapy: At least 4 weeks since the completion of any type of immunotherapy, e.g. tumor vaccines, CAR-T cells, anti-GD2 Monoclonal antibodies (ex. naxitamab, dinutuximab, etc.).
   4. Radiotherapy: At least 30 days since the last treatment except for radiation delivered with palliative intent to a non-target site.
   5. Stem Cell Transplant:

      * Allogeneic: No evidence of active graft vs. host disease
      * Allogeneic/Autologous: ≥ 2 months must have elapsed since transplant.
   6. MIBG Therapy: At least 6 weeks since treatment with MIBG therapy.
7. Subjects must have a Lansky or Karnofsky Performance Scale score of >/= 50.
8. Subjects must have adequate organ function at the time of enrollment:

   * Cardiac: Subjects must have a QTcF ≤ 480 msc.
   * Hematological: Hematological recovery as defined by ANC ≥750/μL
   * Liver: Adequate liver function as defined by AST and ALT <5x upper limit of normal
   * Renal: Subjects must have adequate renal function defined as an estimated Glomerular Filtration rate (eGFR) as calculated from the Bedside Schwartz equation (in units of mL/min/1.73 m2) or via radioisotope GFR ≥ 70.

   The Bedside Schwartz equation is: [(0.413) X (Height in cm)] / SCr
9. Subjects of childbearing potential must have a negative serum pregnancy test. Subjects of childbearing potential must agree to use effective measures to avoid pregnancy.
10. Written informed consent in accordance with institutional and FDA guidelines must be obtained from all subjects (or subjects' legal representative).

Exclusion Criteria:

1. Investigational Drugs: Subjects who are currently receiving another investigational drug are excluded from participation.
2. Anti-cancer Agents: Subjects who are currently receiving other anticancer agents are not eligible. Subjects must have fully recovered from the hematological and bone marrow suppression effects of prior therapy.
3. Subjects who are currently receiving Vitamin K antagonists (warfarin).
4. Subjects who are currently receiving the class of lipid-lowering medications HMG-CoA reductase inhibitors (statins).
5. Infection: Subjects who have an uncontrolled infection are not eligible until the infection is judged to be well controlled in the opinion of the investigator.
6. Subjects who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study, or in whom compliance is likely to be suboptimal, should be excluded.
7. Subjects with any clinically significant unrelated systemic illness (serious infections or significant cardiac, pulmonary, hepatic or other organ dysfunction), that in the opinion of the investigator would compromise the subject's ability to tolerate protocol therapy, put them at additional risk for toxicity or would interfere with the study procedures or results.
8. Subjects with any of the following gastrointestinal disorders:

   1. Active malabsorption (e.g. short gut) syndrome.
   2. Uncontrolled diarrhea (excess of 4 stools/day)
   3. Gastritis, ulcerative colitis, Chron's disease or hemorrhagic coloproctitis
   4. History of gastric or small bowel surgery involving any extent of gastric or small bowel resection
9. Lactating subjects are not eligible unless they have agreed to not breastfeed their infants. There is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the nursing subject with silmitasertib. (NOTE: breast milk cannot be stored for future use while the nursing subject is being treated on study.)
10. Subjects with a history of any other malignancy.

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 104 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2030-11-01 (Estimated); Study Completion 2035-11-01 (Estimated)

PRIMARY OUTCOMES:
Phase I- Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 2 years plus 30 days
  To characterize the safety profile of silmitasertib in combination with chemotherapy
Phase I- Number of Participants with Dose Limiting Toxicities to determine RP2D | 21 days
  To determine the Recommended Phase 2 Dose (RP2D) of silmitasertib in combination with chemotherapy
Phase II- Determine the Overall Response Rate (ORR) of Participants using INRC | 2 years
  To evaluate the efficacy of silmitasertib in combination with chemotherapy in 2 disease cohorts, based upon Overall response rate (ORR)

SECONDARY OUTCOMES:
Phase I- Determine the Overall Response Rate (ORR) of Participants using INRC | 2 years
  To evaluate the efficacy of silmitasertib in combination with chemotherapy in 2 disease cohorts based upon Overall response rate (ORR)
Number of participants with progression free survival (PFS) during study | 2 years
  To evaluate the efficacy of silmitasertib in combination with chemotherapy in 2 disease cohorts based upon Progression Free Survival (PFS)
Phase II- Length of time that participants experience Overall Survival (OS) | 7 years
  To evaluate the efficacy of silmitasertib in combination with chemotherapy in 2 disease cohorts based upon Overall Survival (OS)
Phase II- Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 2 years plus 30 days
  To characterize the safety profile of silmitasertib in combination with chemotherapy
Phase II - Determine the Disease Control Rate (DCR) of participants based on response | 2 years plus 30 days
  Disease Control Rate (DCR): Defined as CR + PR + MR + SD for Neuroblastoma (INRC) and CR + PR + SD for Ewing Sarcoma (RECIST v1.1).

CONTACTS AND LOCATIONS:
Overall Officials: Chandrika Behura, MD, Study Chair — Penn State Health Children's Hospital
Locations (18):
- United States (17):
  - University of Alabama/Children's of Alabama, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Rady Children's Hospital, San Diego, California
  - University of Florida, Gainesville, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - St. Joseph's Children's Hospital, Tampa, Florida
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Norton Children's Research Institute/Affiliated with University of Louisville School of Medicine, Louisville, Kentucky
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Penn State Milton S. Hershey Medical Center and Children's Hospital, Hershey, Pennsylvania
  - Hasbro Children's Hospital, Providence, Rhode Island
  - Monroe Carrell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Children's Medical Center, Dallas, Texas
  - Virginia Commonwealth University, Richmond, Virginia
- UHC Sainte-Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Beat Childhood Cancer Research Consortium website — https://research.beatcc.org/